CLINICAL TRIAL: NCT05527236
Title: The Effect of Breathing Exercises and Virtual Reality Applications During Pregnancy and Labor on Labor Pain, Duration, and Birth Satisfaction: A Randomized Controlled Study
Brief Title: The Effects of Breathing Exercises and Virtual Reality Applications During Pregnancy and Labor.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semra Çevik, phD (Other)
Responsible Party: Sponsor-Investigator, Semra Çevik, phD, Associate Professor, University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Virtual Breathing
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Labor Pain; Labor Onset; Patient Satisfaction; Virtual Reality; Breathing; Tic
Keywords: breathing exercises; virtual reality; pain intensity; duration of labor; birth satisfaction
MeSH Terms: conditions — Labor Pain; Patient Satisfaction; Respiratory Aspiration; Tics; Pain | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breathing Exercise Group (Experimental): The research was carried out in two stages. In the first stage, for the experimental groups at the 36th-39th weeks of pregnancy, a 10-minute breathing exercise was performed 3 times a week using virtual reality glasses and a breathing exercise device. In the second stage of the study (when the cervical dilatation was 4 cm), the breathing exercise group was made breathing exercise again. As soon as the virtual reality glasses and breathing exercise device were removed, VAS was applied. In order to evaluate the second and third stages of labor, the birth evaluation section of the labor observation form was filled out. Satisfaction with birth was evaluated with the ''Birth Satisfaction Scale'' within the first 4 hours after birth after the delivery was completed.
  Interventions: Other: Breathing Exercise
- Virtual Reality Group (Experimental): The research was carried out in two stages. In the first stage, for the experimental groups at the 36th-39th weeks of pregnancy, a 10-minute breathing exercise was performed 3 times a week using virtual reality glasses and a breathing exercise device. In the second stage of the study (when the cervical dilatation was 4 cm), the virtual reality group watched a 10-minute video with virtual reality glasses. Once the virtual reality glasses were removed from experimental groups Visual Analogue Scale was applied. Birth satisfaction was evaluated with the Birth Satisfaction Scale within the first 4 hours after the delivery was completed.
  Interventions: Other: Virtual Reality
- Control Group (No Intervention): Descriptive information form was filled out at 36th week of pregnancy in a quiet pregnant outpatient clinic in the hospital. After participants were admitted to the delivery room of Gaziantep Cengiz Gökçek Obstetrics and Pediatrics Hospital at the 40th week of pregnancy, and taken to their beds, in labour observation form, the labour section and the birth evaluation section which is used to evaluate the second and third stages of labour were filled out. Then, VAS was applied when cervical dilatation was 4 cm (the beginning of the active phase). Birth satisfaction was evaluated with the ''Birth Satisfaction Scale'' within the first 4 hours after birth after the delivery was completed.
  No application was made to pregnant women in this group, except for routine practices in the pregnant outpatient clinic at the hospital and in the delivery room.

INTERVENTIONS:
Other: Breathing Exercise — The research was carried out in two stages. In the first stage, for the experimental groups at the 36th-39th weeks of pregnancy, a 10-minute breathing exercise was performed 3 times a week using virtual reality glasses and a breathing exercise device. In the second stage of the study (when the cervical dilatation was 4 cm), the breathing exercise group was made breathing exercises again. As soon as the virtual reality glasses and breathing exercise device were removed, VAS was applied. In order to evaluate the second and third stages of labor, the birth evaluation section of the labor observation form was filled out. Satisfaction with birth was evaluated with the ''Birth Satisfaction Scale'' within the first 4 hours after birth after the delivery was completed.
  Arms: Breathing Exercise Group
Other: Virtual Reality — The research was carried out in two stages. In the first stage, for the experimental groups at the 36th-39th weeks of pregnancy, a 10-minute breathing exercise was performed 3 times a week using virtual reality glasses and a breathing exercise device. In the second stage of the study (when the cervical dilatation was 4 cm) the virtual reality group watched a 10-minute video with virtual reality glasses. Once the virtual reality glasses were removed from experimental groups Visual Analogue Scale was applied. Birth satisfaction was evaluated with the Birth Satisfaction Scale within the first 4 hours after the delivery was completed.
  Arms: Virtual Reality Group

SUMMARY:
Aim and Objectives: The purpose of this study was to determine the effects of breathing exercises and virtual reality applications during pregnancy and labor on labor pain, duration, and birth satisfaction.

Background: Conducted studies show that practices such as virtual reality have positive effects on labor. However, there is no study that compares the effects of breathing exercises with virtual reality applications on labor.

Design: A randomized controlled experiment was conducted by the CONSORT guidelines.

Methods: The study included 114 pregnant women (Breathing Exercise Group:39, Virtual Reality Group:37, Control Group:38). The research was carried out in two stages. In the first stage, for the experimental groups at the 36th-39th weeks of pregnancy, a 10-minute breathing exercise was performed 3 times a week using virtual reality glasses and a breathing exercise device. In the second stage of the study (when the cervical dilatation was 4 cm), the breathing exercise group was made breathing exercises again. The virtual reality group watched a 10-minute video with virtual reality glasses. Once the virtual reality glasses were removed from experimental groups Visual Analogue Scale was applied. Birth satisfaction was evaluated with the Birth Satisfaction Scale within the first 4 hours after the delivery was completed.

DETAILED DESCRIPTION:
1. INTRODUCTION Management of labor pain and increasing the birth satisfaction level of the expectant mother are the main goals of prenatal and postpartum care (Huntley, Coon, & Ernest, 2004). For this purpose, two kinds of methods, which are pharmacological and non-pharmacological are used (Vulkan, & Yıldız, 2016).

   One of the non-pharmacological applications is virtual reality technology (Dockx et al., 2016; Ebrahimian, & Bilandi, 2022).

   Another non-pharmacological application in pregnancy and labor is breathing exercises (Dikmen, & Sanlı, 2019).
2. MATERIAL AND METHODS Study design The researchers carried out this study between October 2020 and January 2022 in the pregnant outpatient clinic and in the delivery room, at the maternity hospital in southeastern Anatolia, Turkey.

Study population The sample of the study consisted of all pregnant women who applied to the pregnancy polyclinic for normal delivery. The sample size of the study was calculated as 63 pregnant women including 21 participants in each group using the G*Power Software version 3.9.1 with the VAS mean scores in the study by Dutucu (2019) as 5.63 (SD = 1.07), and obtaining a rate of 80% in the power test, an alpha value of 0.05 with a 95% confidence level (Dutucu, 2019). However, we decided to include 40 pregnant women in each group in order to be able to generalize and strengthen the research results. The study reached 120 pregnant women. Five pregnant women did not meet the inclusion criteria and one pregnant woman withdraw from the study during the process and was excluded from the study. Eventually, the study sample was composed of 114 pregnant women based on the CONSORT 2010 flow diagram: 39 in the breathing exercise group, 37 participants in the virtual reality group, and 38 in the control group.

Randomization Pregnant women were randomly selected via a drawing, and they were assigned to either the experimental or control group. For the drawing of lots; 120 small papers were prepared, and the words 'virtual', 'breathing', and 'control' were written on every 40 papers, and they were folded and put into a bag. The inclusion of pregnant into groups was determined according to the papers pregnant drew from the bag. Pregnant women participating in the study did not know how many groups are available and which method will be applied to the group in which they are selected. We carried out this study with three groups, one control, and two experiments. The experimental group is divided into two groups, the breathing exercise group, and the virtual reality group.

Data Collection Tools The data of the study were collected by using "Descriptive Information Form", "Labour Observation Form", "Visual Analog Scale ", and "Birth Satisfaction Scale".

Collection of data The First Stage of The Research As mentioned before, this step was applied in the same way for both experimental groups. The descriptive information form was filled in by the pregnant women under the supervision of the researchers. At the 36th gestational week, the pregnant women were informed that they should not eat or drink anything 1 hour before the exercise. In addition, we gave the necessary information to the participants about virtual reality and breathing exercise devices together with how they would be applied and what video content they would watch. A 10-minute(5 minutes of breathing exercise and 5 minutes of relaxation exercise at the end of the exercise) breathing exercise video was shown to the participants using virtual reality glasses. At the same time, the participants were asked to do the breathing exercises shown in the video using the breathing exercise device. This application was performed 3 times a week from the 36th gestational week to the 40th gestational week, and 12 times in total until birth.

All applications were carried out in a quiet, calm pregnant outpatient clinic in the hospital, and a cushion on which the pregnant woman could sit and a pillow that could support her back were used to ensure the comfort of the pregnant woman.

The Second Stage of The Research After the first stage of the research was applied to the experimental groups, the second stage was carried out during the delivery at the 40th week of pregnancy. The second stage was applied in a different way for the Breathing Exercise Group and Virtual Reality Group. In the following sections, the second stage is explained for both groups.

Breathing Exercise Group Participants after being admitted to the delivery room of Gaziantep Cengiz Gökçek Obstetrics and Pediatrics Hospital and taken to their beds, the labor evaluation section of the labor observation form was filled. Firstly the pregnant women were placed in the semi-fowler position and virtual reality glasses with a breathing exercise device were put on when the cervical dilatation was 4 cm (the beginning of the active phase). A 10-minute (5 minutes of breathing exercise and 5 minutes of relaxation exercise at the end of the exercise) breathing exercise video was shown to the participants using virtual reality glasses. At the same time, the participants were asked to do the breathing exercises shown in the video using the breathing exercise device. As soon as the virtual reality glasses and breathing exercise device were removed, VAS was applied. In order to evaluate the second and third stages of labor, the birth evaluation section of the labor observation form was filled out. Satisfaction with birth was evaluated with the ''Birth Satisfaction Scale'' within the first 4 hours after birth after the delivery was completed.

Virtual Reality Group Participants after being admitted to the delivery room of Gaziantep Cengiz Gökçek Obstetrics and Pediatrics Hospital and taken to their beds, the labor evaluation section of the labor observation form was filled. Firstly the pregnant women were placed in the semi-fowler position and virtual reality glasses were put on when the cervical dilatation was 4 cm (the beginning of the active phase). Then, in virtual reality glasses, a 10-minute relaxing video of the chirping of birds, calm sea, colorful birds, sunrise, sunset, colorful flowers, and trees was played accompanied by the background music called ''Dancing With Nature'' by Tim Janis. Once the virtual reality glasses were removed VAS was applied. In order to evaluate the second and third stages of labor, the birth evaluation part of the labor observation form was filled out. Birth satisfaction was evaluated with the ''Birth Satisfaction Scale'' within the first 4 hours after the delivery was completed.

Control Group A descriptive information form was filled out at the 36th week of pregnancy in a quiet pregnant outpatient clinic in the hospital. After participants were admitted to the delivery room of Gaziantep Cengiz Gökçek Obstetrics and Pediatrics Hospital at the 40th week of pregnancy, and taken to their beds, in labor observation form, the labor section and the birth evaluation section which are used to evaluate the second and third stages of labor were filled out. Then, VAS was applied when cervical dilatation was 4 cm (the beginning of the active phase). Birth satisfaction was evaluated with the ''Birth Satisfaction Scale'' within the first 4 hours after birth after the delivery was completed.

No application was made to pregnant women in this group, except for routine practices in the pregnant outpatient clinic at the hospital and in the delivery room.

ELIGIBILITY:
Inclusion Criteria:

* In the 36th week of pregnancy,
* Those who gave birth at 40 weeks of gestation,
* Those who will have a normal (vaginal) birth,
* Primiparas,
* 19 years old and over,
* Able to communicate verbally,
* Who agreed to participate in the study,
* Those who can read and write,
* Those who have COVID-19 test negative, no contact or doubt.

Exclusion Criteria:

* Have no risks regarding the pregnant woman and fetus,
* Multiparous,
* Those who underwent cesarean section,
* Having visual or auditory impairment,
* Having any infection in the mouth,
* Having any contagious eye disease,
* Those administered analgesics during labour,
* Those who have COVID-19 test positive, contact or doubt.

Ages: 19 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
''Labor pain'' | ''1 minute later''
  Labor pain was evaluated with the Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
''Duration of labor'' | ''within the first 10 hours''
  Duration of labor was evaluated with the Labour Observation Form.
''Birth satisfaction'' | ''within the first 4 hours''
  Birth satisfaction was evaluated with the Birth Satisfaction Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Cengiz Gökçek Obstetrics and Pediatrics Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No